CLINICAL TRIAL: NCT02617043
Title: Hypofractionated Whole-breast Irradiation With Simultaneously Integrated Boost For Early-Stage Breast Cancer After Breast-conserving Surgery
Acronym: HF-WBI-SIB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoli Yu, Associate Professor of department of radiation oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-BC001
Record Dates: First submitted 2015-11-19; First posted 2015-11-30 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; hypofractionated whole breast irradiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HF-WBI (Experimental): Hypofractionated whole breast irradiation for early breast cancer with prescription dose 40Gy in 15 fractions in 3 weeks. Tumor bed is simultaneously integrated boosted to 48Gy.
  Interventions: Radiation: hypofractionated whole breast irradiation with simultaneously integrated boost

INTERVENTIONS:
Radiation: hypofractionated whole breast irradiation with simultaneously integrated boost — deliver 40Gy/15Fx to whole breast with 48Gy/15fx simultaneously integrated to tumor bed

SUMMARY:
The study was designed to evaluate the feasibility and safety of hypofractionated whole-breast irradiation with simultaneously integrated boost for early-stage breast cancer after breast conserving surgery in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-60 years old
* Treated with breast conversing surgery and sentinel lymph node biopsy or axillary lymph node dissection
* Pathologically confirmed invasive breast cancer
* A pathological T1-2N0M0 tumor
* Tumor bed is labeled with Titanium clips
* Negative surgical margins
* Written informed consent.

Exclusion Criteria:

* KPS<70
* Treated with neoadjuvant chemotherapy
* Sentinel lymph nodes only containing isolated tumour cells (<0.2 mm)
* With severe comorbidity
* Previous breast cancer or other malignant tumor history
* Previous radiotherapy for breast or thorax
* Medical contraindication for radiotherapy
* Pregnant or nursing

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with treatment-related toxicity assessed by CTCAE v4.0 | 2 year
  acute toxicity related to irradiation such as lung and skin

SECONDARY OUTCOMES:
acute radiation-induced toxicity assessed by CTCAE v4.0 | during radiotherapy; 3months; 6 months
  acute toxicity related to skin and lung
local-regional recurrence | 5 years
Disease free survival | 5 years
Overall survival Over survival | 5 years
Late complications | 1,2,3,4,5years
cosmetic effect measured by Harvard 4 scale evaluation system | 2,3,4,5years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Yu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China